CLINICAL TRIAL: NCT01222026
Title: Primary Hyperparathyroidism: Does a Systematic Treatment Improve the Calcium- and Bone Metabolism After Successful Surgery? - Part I
Brief Title: Systematic Treatment After Successful Surgical Treatment for Primary Hyperparathyroidism With Strontium Ranelate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Martin Niederle, MD, PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK Nr 214/2008; 2008-001703-32 (EudraCT Number)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Primary Hyperparathyroidism; Osteopenia; Osteoporosis
Keywords: Primary Hyperparathyroidism; Osteopenia; Osteoporosis
MeSH Terms: conditions — Hyperparathyroidism, Primary; Bone Diseases, Metabolic; Osteoporosis | interventions — strontium ranelate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strontium Ranelate (Active Comparator): Receiving Strontium Ranelate + Ca/Vitamin-D
  Interventions: Drug: Strontium Ranelate + Ca/Vitamin-D
- Placebo (Placebo Comparator): Receiving Placebo + Ca/Vitamin D
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Strontium Ranelate + Ca/Vitamin-D — 2g Strontium Ranelate once daily 1000mg Calcium 800 IE Vitamin D
  Other Names: Protelos (r)
  Arms: Strontium Ranelate
Drug: Placebo — Placebo 1000mg Calcium 800 IE Vitamin-D
  Arms: Placebo

SUMMARY:
Patients with primary hyperparathyroidism (pHPT) with osteopenia and osteoporosis are treated with strontium ranelate/Ca+Vitamin-D or placebo/Ca+Vitamin D after successful surgical treatment of pHPT.

Strontium ranelate/Ca + Vitamin-D helps to regain bone mass in patients with osteopenia or osteoporosis after successful parathyroidectomy for pHPT and results in higher gain of BMD than placebo treated patients.

DETAILED DESCRIPTION:
The chronic excessive hypersecretion of parathyroid hormone (PTH) has significant impact on bone remodeling. In primary hyperparathyroidism (PHPT) bone turnover is increased, resulting in a higher resorption of bone and thus loss of bone density.

After successful surgical treatment of pHPT bone metabolism switches from catabolic state to anabolic state again. However studies show that especially postmenopausal women regain significantly less BMD but these women suffer from osteopenia and osteoporosis most often and would need to regain as much bone mass as possible to prevent fractures. The optimal state would be to reach normal BMD again. Although this state is hardly reachable especially these patients may benefit from a treatment acting anti-resorptive and rising bone formation. The only drug combining these qualities known so far is Strontium ranelate.

Therefore the hypothesis is that Strontium ranelate/Ca + Vitamin-D helps to regain bone mass in patients with osteopenia or osteoporosis after successful parathyroidectomy for pHPT and results in higher gain of BMD than placebo treated patients.

ELIGIBILITY:
Inclusion Criteria:

* biochemically proven PHPT, PTX planned
* osteopenia (t-score < -1 and > -2.5) or osteoporosis (t-score ≤ -2.5) according to WHO Criteria [27]

Exclusion Criteria:

* Premenopausal women
* Cancer (lung, breast, prostatic, parathyroid cancer and thyroid carcinoma >1cm)
* Persisting or recurrent PHPT (postoperative hypercalcemia)
* Four-gland hyperplasia
* Multiple endocrine neoplasia (MEN) or hereditary PHPT
* Familial hypocalciuric hypercalcaemia (Ca/creatinine ratio < 0.01)
* Anamnestic pulmonal embolism or deep venous thrombosis
* Blood coagulation disorder or coagulopathy
* Phenylketonuria
* Renal impairment (creatinine clearance <30ml/h)
* Severe hepatic disorder
* Severe systemic disorder
* Thyroid dysfunction
* Immobilisation
* Intake of drugs with potential effects on BMD like glucocorticoids, lithium, estrogen-replacement therapy, selective Estrogen-receptor modulators (sERMs), bisphosphonates in the last three months
* Known allergy against any component of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density measurement of the Lumbar spine | 1 year

SECONDARY OUTCOMES:
Bone mineral density of the femoral neck | 1 year
Bone mineral density of the radius | 1 year
Osteoprotegerin (OPG/OCIF) | 1 year
RANKL (OPG-ligand) | 1 year
cathepsin K (cat K) | 1 year
ionised calcium (Ca++) | 1 year
phosphate (PO4-) | 1 year
alkaline phosphatase (AP) | 1 year
bone-specific alkaline phosphatase (BAP) | 1 year
osteocalcin (Oc) | 1 year
parathyroid hormone (PTH) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Niederle, Prof., MD, Principal Investigator — Section of Endocrine Surgery, Department of Surgery, Medical University of Vienna
Locations (1):
- Medical University Vienna, General Hospital Vienna (AKH Wien), Vienna, Vienna, Austria